CLINICAL TRIAL: NCT02388009
Title: Safety and Tolerability of a Candidate Bioconjugate Vaccine Against Shigella Flexneri 2a When Administered to Adult Volunteers
Brief Title: Safety and Tolerability of a Bioconjugate Vaccine Against Shigella Flexneri 2a
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LimmaTech Biologics AG (Industry)
Collaborators: Wellcome Trust (Other); Naval Medical Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SF2A-1
Record Dates: First submitted 2015-02-23; First posted 2015-03-13 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Shigellosis
Keywords: bioconjugate vaccine; safety; immunogenicity; shigellosis
MeSH Terms: conditions — Dysentery, Bacillary | interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Flexyn2a (Active Comparator): 2 doses of 10 μg of Flexyn2a will be injected intramuscularly 4 weeks apart
  Interventions: Biological: Flexyn2a
- Flexyn2a plus adjuvant (Active Comparator): 2 doses of 10 μg of Flexyn2a plus adjuvant will be injected intramuscularly 4 weeks apart
  Interventions: Biological: Flexyn2a plus adjuvant
- Placebo (Placebo Comparator): 2 doses of saline buffer plus adjuvant will be injected intramuscularly 4 weeks apart
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Flexyn2a — Intramuscular doses of 0.5 mL
  Arms: Flexyn2a
Biological: Placebo — Intramuscular doses of 0.5 mL
  Arms: Placebo
Biological: Flexyn2a plus adjuvant — Intramuscular doses of 0.5 mL
  Arms: Flexyn2a plus adjuvant

SUMMARY:
This is a phase I, single-blind, randomized, placebo-controlled, single-center study in healthy subjects using a staggered approach to dosing.

30 subjects will be randomized to receive 10 μg Flexyn2a candidate vaccine with or without adjuvant or placebo.

DETAILED DESCRIPTION:
A total of 30 subjects will be randomly assigned to one of 3 different arms in order to evaluate the safety, tolerability and immunogenicity of a candidate vaccine, formulated with or without adjuvant, and the outcome compared to a placebo control group.

For each active treatment group, 12 subjects will be injected twice with 10 μg Flexyn2a candidate vaccine 4 weeks apart. A control group with 6 subjects will be injected following the same schedule with a placebo solution.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female volunteers, age of 18 to 50 years (inclusive) at the time of enrollment.
2. Signed informed consent form.
3. Completion and review of comprehension test (achieved >70% accuracy)
4. Available for the required follow-up period and scheduled clinic visits.
5. Women: negative pregnancy test with understanding (through informed consent process) to not become pregnant or or breastfeed during the study or within twelve (12) weeks after the last vaccine dose.

Exclusion Criteria:

1. Health condition that, in the opinion of the investigator, may interfere with optimal participation in the study or place the volunteer at increased risk of adverse Events (AEs). Study clinicians, in consultation with the PI, will use clinical judgment on a case by-case basis to assess safety risks under this criterion. The PI will consult with the Research Monitor as appropriate.
2. Clinically significant abnormalities on physical examination.
3. Clinically significant abnormalities on basic laboratory screening.
4. Presence of significant unexplained laboratory abnormalities that, in the opinion of the PI, may potentially confound the analysis of the study results
5. Regular use of constipation, antacid or anti-diarrheal medications or treatments.
6. Abnormal stool pattern (fewer than 3 stools per week or more than 3 per day) or loose/liquid stools more than occasionally.
7. Use of immunosuppressive drugs such as corticosteroids or chemotherapeutics that may influence antibody development.
8. Women currently nursing.
9. Participation in research involving another investigational product (defined as receipt of investigational product or exposure to invasive investigational device) within 30 days of planned date of first vaccination or anytime throughout the duration of the study.
10. Positive blood test for HBsAg, hepatitis C Virus (HCV), HIV-1.
11. Positive blood test for HLA-B27.
12. Immunosuppressive illness or immunoglobulin deficiency (serum immunoglobulin A level < 7 mg/dL or limit of detection of assay).
13. Family history of congenital or hereditary immunodeficiency.
14. Treatment with immunoglobulins or blood products within 3 months from first candidate vaccine injection.
15. History of microbiologically confirmed Shigella infection.
16. Personal or family history of inflammatory arthritis.
17. Personal or family history of irritable bowel syndrome.
18. Received previous experimental Shigella vaccine or live Shigella challenge.
19. Have had diarrhea while traveling outside the United States or lived for 2 or more months during the past 3 years in a country with potentially higher Shigella infection rates, including Africa, South America, Central America, and Asia (except Japan).
20. Occupation involving handling of Shigella bacteria currently, or in the past 3 years.
21. History of allergy to any vaccine.
22. History of allergy to aluminum hydroxide.
23. Serum immunoglobulin G endpoint titer ≥ 2500 to Shigella Lipopolysaccharide.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-02; Primary Completion 2015-05 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Occurrence and severity of adverse events | until Day 56
  Number and severity of local site injection and general adverse events will be collected and compared between the different arms of the study

SECONDARY OUTCOMES:
Evaluation of antigen-specific antibodies between baseline (D0) and after injection for all groups. | until Day 56
  Immunogenicity will be evaluated after the first and second injection and compared to pre-immune levels
Evaluation of antigen-specific antibodies between subjects receiving the candidate vaccine with and without adjuvant | until Day 56
  Immunogenicity will be compared between subjects receiving candidate vaccine with and without adjuvant after the first and second injection

CONTACTS AND LOCATIONS:
Overall Officials: Mark S. Riddle, MD Dr Ph, Principal Investigator — Navy Medical Research Center
Locations (1):
- WRAIR Clinical Trial Center (CTC), Silver Spring, Maryland, United States

REFERENCES:
- [Derived] Riddle MS, Kaminski RW, Di Paolo C, Porter CK, Gutierrez RL, Clarkson KA, Weerts HE, Duplessis C, Castellano A, Alaimo C, Paolino K, Gormley R, Gambillara Fonck V. Safety and Immunogenicity of a Candidate Bioconjugate Vaccine against Shigella flexneri 2a Administered to Healthy Adults: a Single-Blind, Randomized Phase I Study. Clin Vaccine Immunol. 2016 Dec 5;23(12):908-917. doi: 10.1128/CVI.00224-16. Print 2016 Dec. PMID 27581434